CLINICAL TRIAL: NCT02187133
Title: A Phase Ib Dose Escalation Trial of Carfilzomib in Combination With Bendamustine and Rituximab In Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Carfilzomib With Bendamustine and Rituximab in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, C. Babis Andreadis, Associate Professor of Clinical Medicine, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14251; NCI-2015-00775 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Recurrence | interventions — carfilzomib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receive carfilzomib IV over 30 minutes twice weekly on days 1, 2, 8, 9, 15, and 16 or weekly on days 2, 9, and 16; bendamustine hydrochloride IV over 60 minutes on days 1 and 2; and rituximab IV over 30-90 minutes on day 9 (course 1 only) and day 1 (subsequent courses). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Carfilzomib — Given IV; Dose Level (DL)
  Twice Weekly:
  DL -1 and DL 1: 15 mg/m^2
  Weekly:
  DL 1.5: 20,27,27 mg/m^2, DL 2: 20,36,36 mg/m^2, DL 3: 20,56,56 mg/m^2 DL 4: 20,70,70 mg/m^2
  Other Names: Kyprolis; PR-171
Drug: Bendamustine — Given IV; Dose Level (DL)
  DL -1: 75 mg/m^2 DL 1,1.5, 2, 3, and 4: 90 mg/m^2
  Other Names: Bendamustine Hydrochloride; Cytostasan Hydrochloride; Levacet; Ribomustin; Treanda
Drug: Rituximab — Given IV; 375 mg/m^2
  Other Names: C2B8 Monoclonal Antibody; Rituxan; RTXM83

SUMMARY:
This study will be conducted as a Phase Ib, open-label, non-randomized, single-institution study to evaluate the safety and tolerability of carfilzomib in combination with bendamustine and rituximab in patients with relapsed or refractory NHL and to determine the recommended phase II dose and preliminary efficacy of this combination. The study will have two phases: a dose-escalation phase to determine the maximal tolerated dose of carfilzomib in this combination where participants will be monitored for toxicity, tolerability and response and a dose-expansion phase that will determine the preliminary efficacy in patients with Mantle cell lymphoma or any other disease subtype in which there is a preliminary efficacy signal observed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of carfilzomib when combined with bendamustine (bendamustine hydrochloride) and rituximab in patients with relapsed or refractory non-Hodgkin's lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary antitumor activity of carfilzomib with bendamustine and rituximab in patients with non-Hodgkin lymphoma (dose escalation) and with specific non-Hodgkin lymphoma (NHL) subtypes (dose expansion).

OUTLINE: This is a dose-escalation study of carfilzomib.

Patients receive carfilzomib intravenously (IV) over 30 minutes twice weekly on days 1, 2, 8, 9, 15, and 16 or weekly on days 2, 9, and 16; bendamustine hydrochloride IV over 60 minutes on days 1 and 2; and rituximab IV over 30-90 minutes on day 9 (course 1 only) and day 1 (subsequent courses). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks for 6 months, every 3 months for 6 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed B-cell non-Hodgkin's lymphoma (Mantle Cell Lymphoma, Follicular Lymphoma, Small Lymphocytic Lymphoma/Chronic Lymphocytic Leukemia, Marginal Zone Lymphoma, Diffuse Large B-cell Lymphoma, and Lymphoplasmacytic Lymphoma)
* Must have relapsed or refractory disease after 2 or more prior lines of therapy; 1 line of therapy is allowed, if it included an autologous stem cell transplant and at least 12 weeks have elapsed from Day 0. A line of therapy is defined as a course of therapy that is not interrupted by progressive disease.
* Subjects must have measurable disease of at least 1.5 cm in diameter
* Age ≥ 18 years
* Life expectancy ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception. FCBP definition: A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months.
* Male subjects must agree to practice contraception for at least 90 days after the last dose of carfilzomib, and must agree not to donate sperm for at least 90 days after the last dose of carfilzomib

Adequate bone marrow function:

* Absolute neutrophil count ≥ 1.0 × 10^9/L
* Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior Cycle 1, Day 1 (subjects may be receiving red blood cell (RBC) transfusions in accordance with institutional guidelines)
* Platelet count ≥ 75 × 10^9/L or≥ 50× 10^9/L if there is lymphoma involvement in the bone marrow, independent of platelet transfusion

Adequate hepatic function:

* Serum aspartate aminotransferase (AST) /alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal
* Serum direct bilirubin ≤ 2 mg/dL (unless history of Gilbert's)

Adequate renal function:

* Creatinine clearance (CrCl) ≥ 30 mL/minute, either measured or calculated using a standard formula (eg, Cockcroft and Gault)
* Uric acid If elevated, corrected to within laboratory range prior to dosing

Exclusion Criteria:

* Progressive disease on bendamustine within 6 months of cycle 1, Day 1
* Prior treatment with carfilzomib for lymphoma
* Patient has received other investigational drugs within 21 days prior to Cycle 1, Day 1. Exceptions allowed if greater than four half-lives of the experimental agent ).
* Prior radiation therapy or chemotherapy within 2 weeks prior Cycle 1, Day 1, monoclonal antibody therapy within 4 weeks
* Prior allogeneic transplant
* Active, uncontrolled central nervous system (CNS) involvement by lymphoma
* Pregnant or lactating females
* Major surgery within 14 days prior Cycle 1, Day 1
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior Cycle 1, Day 1
* Known human immunodeficiency virus infection
* Active hepatitis C infection (HCV), defined as presence of HCV antibody.
* Unstable angina or myocardial infarction within 6 months prior Cycle 1, Day 1, New York Heart Association (NYHA) Class III or IV heart failure, left ventricular ejection fraction (LVEF) < 40%, uncontrolled angina, history of severe coronary artery disease, history of torsade de pointes, history of symptomatic pulmonary hypertension, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, QTc prolongation >450 msec, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior Cycle 1, Day 1
* Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior Cycle 1, Day 1
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior Cycle 1, Day 1
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) | Up to 1 cycle (28 days per cycle)
  The MTD will be the dose level immediately preceding the dose level at which >= 2 Dose Limiting Toxicities (DLT) are observed and at which 0/3 or 1/6 participants experiences a DLT.
Number of participants with Dose Limiting Toxicities (DLT) | Up to 1 cycle (28 days per cycle)
  The DLT period will correspond to cycle 1 of therapy. The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 will be used to assess the severity of adverse events. The causality of each AE will be assessed by the investigator for confirmation of a DLT.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  The lymphoma response assessment will be determined using the revised International Working Group (IWG) criteria for Complete Response (CR) defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy, a post-treatment residual mass of any size is permitted as long as it is Positron Emission Tomography (PET) negative, the spleen and/or liver, if enlarged before therapy on the basis of the physical examination or CT scan, should not be palpable on physical examination and should be considered normal size by imaging studies, and nodules related to lymphoma should disappear, etc. or Partial Response (PR) defined as the post-treatment PET should be positive in at least one previously involved site, At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses, No new sites of disease should be observed, etc.
Median Duration of Response | Up to 2 years
  Defined as the time from documentation of PR or CR until documented lymphoma progression or receipt of anti-lymphoma therapy or death due to lymphoma. Patients are to be censored at the time of last follow-up or death due to another cause.
Median Progression Free Survival (PFS) | Up to 2 years
  Defined as the time from day 1 until lymphoma progression, receipt of anti-lymphoma therapy, or death as a result of any cause. Patients will be censored at the time of last follow up.
Median Time to Next Therapy | Up to 2 years
  Time to next therapy is measured from day 1 to receipt of anti-lymphoma therapy or death due to lymphoma. Patients are censored at the time of last follow-up or death unrelated to treatment or disease.

OTHER OUTCOMES:
Median Overall Survival | Up to 2 years
  Defined as the time from day 1 until death as a result of any cause. Patients will be censored at the time of last follow-up
Correlation of antitumor activity with markers of activation of the terminal unfolded protein response (UPR) or modulation of the apoptotic pathway in primary tumor tissue. | Up to 2 years
  The molecular events associated with the terminal UPR and apoptotic pathways will be correlated to assess their predictive utility for response to therapy with carfilzomib in combination with bendamustine.
Correlation of treatment-related toxicity with markers of activation of the terminal unfolded protein response (UPR) or modulation of the apoptotic pathway in primary tumor tissue. | Up to 2 years
  The molecular events associated with the terminal UPR and apoptotic pathways will be correlated to assess their predictive utility for response to toxicity with carfilzomib in combination with bendamustine.

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Andreadis, M.D., Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kambhampati S, Fakhri B, Ai WZ, Kaplan LD, Tuscano JM, Wieduwilt MJ, Sudhindra A, Cavallone E, Reiner J, Aoun C, Castillo M, Martinelli M, Ta T, Le D, Padilla M, Crawford E, Andreadis CB. Carfilzomib in Combination With Bendamustine and Rituximab in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma: A Phase I Trial. Clin Lymphoma Myeloma Leuk. 2021 Mar;21(3):139-146. doi: 10.1016/j.clml.2020.12.020. Epub 2020 Dec 24. PMID 33478921